CLINICAL TRIAL: NCT01909674
Title: Differences in Efficacy Between Nasal and Oronasal Masks in the Treatment of Obstructive Sleep Apnea With Continuous Positive Airway Pressure (CPAP): A Randomized Cross-over Study
Brief Title: Differences in Efficacy Between Nasal and Oronasal Masks in the Treatment of OSA With CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1108011845
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oronasal Mask (Experimental): Initial administration of oronasal CPAP mask
  Interventions: Device: Switch CPAP mask type
- Nasal Mask (Experimental): Initial administration of nasal CPAP mask
  Interventions: Device: Switch CPAP mask type

INTERVENTIONS:
Device: Switch CPAP mask type

SUMMARY:
Our group previously conducted a study looking at the performance of three styles of positive airway pressure masks during laboratory treatment studies for obstructive sleep apnea, and we found that patients using a full-mask mask required higher positive airway pressures than patients using nasal or nasal pillows style masks to achieve successful reduction of respiratory events. In the current study we want to randomly assign patients to either nasal or full-face masks and then switch to a different mask (if nasal was originally chosen than the mask will be switched to full-face and vise versa) after 3-weeks of use to see if the number of respiratory events change with the different mask style. We expect the number of respiratory events will increase with the use of full-face masks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* previously diagnosed with OSA
* returning for PAP titrations at the Center for Sleep Medicine
* CPAP and titration naive
* Must have a Apnea/Hypopnea Index (AHI) of ≥ 16/hr.

Exclusion Criteria:

* Patients with ≥ 50% central apneas

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Center for Sleep Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oronasal Mask: Initial administration of oronasal CPAP mask
  Switch CPAP mask type
- Nasal Mask: Initial administration of nasal CPAP mask
  Switch CPAP mask type
Period: Overall Study
Arm/Group | Oronasal Mask | Nasal Mask
Started | 12 | 9
Completed | 7 | 7
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oronasal Mask | Nasal Mask | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 11 | 8 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Effectiveness of Nasal Versus Oronasal CPAP Masks
Description: Total Sleep Time (TST) The amount of actually sleep time in a sleep episode; this time is equal to the total sleep episode less the awake time. TST is the total of all REM and NREM sleep in a sleep episode.
Time Frame: 3 weeks for each mask condition
Population: higher values represent a better outcome
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Total Sleep Time - Nasal Mask; Total Sleep Time (TST) Oronasal Mask: Total Sleep Time (TST)
  The amount of actually sleep time in a sleep episode; this time is equal to the total sleep episode less the awake time. TST is the total of all REM and NREM sleep in a sleep episode.
Arm/Group | Total Sleep Time - Nasal Mask | Total Sleep Time (TST) Oronasal Mask
Number analyzed (Participants) | 7 | 7
minutes | 332.64 (92.09) | 346.79 (86.74)

ADVERSE EVENTS:
Arm/Group | Oronasal Mask | Nasal Mask
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes